CLINICAL TRIAL: NCT02758925
Title: Phase 2 Study of Cytarabine in Association With Bendamustine and Rituximab in the Treatment of Relapsed/Refractory Diffuse Large B Cell Lymphoma
Brief Title: CyBeR Association in Relapsed/Refractory DLBCL
Acronym: CyBeR-Lymph
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Emilie REBOURSIERE, MD, University Hospital, Caen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-005837-37
Record Dates: First submitted 2016-04-14; First posted 2016-05-03 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Bendamustine Hydrochloride; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLBCL patients (Experimental): they will receive a combination of: Rituximab 375mg/m2 IV at Day 1 Bendamustine 90mg/m2 IV at Day 1 and 2 Cytarabine 1000mg/m2 IV at day 2 every 21 days for 6 cycles
  Interventions: Drug: Rituximab; Drug: Bendamustine; Drug: Cytarabine

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 IV day 1
  Other Names: mabthera
Drug: Bendamustine — 90mg/m2 IV day 1-2
  Other Names: levact
Drug: Cytarabine — 1000mg/m2 or 750mg/m2 at day 2 if patients aged more than 70 years or toxicity grade 3/4
  Other Names: aracytine

SUMMARY:
Forty percent of patients with diffuse large B cell lymphoma (DLBCL) have primary refractory or relapsed disease (R/R). For these fit patients, standard treatment in second line therapy is high dose therapy with autologous stem cell transplantation (ASCT). In 48% of DLBCL no ASCT is possible due to progressive disease. For these patients or ineligible to transplantation patients, salvage therapy is often rituximab-gemcitabine-oxaliplatine regimen with an overall response rate (ORR) about 50%.

Bendamustine in combination with rituximab, used as a single agent in the setting of R/R DLBCL patients, have shown an ORR of 62.7% and 45.8% with a good safety profile.

Bendamustine and cytarabine (BAC) showed high synergy in inducing cell death in mantle cell lymphoma and DLBCL cell lines. In a recent phase II study, the combination of cytarabine with Rituximab and Bendamustine (R-BAC) in patients with mantle cell lymphoma who were previously untreated, refractory or relapsed was evaluated.

The efficacy and safety of the R-BAC association will be evaluated in this phase II trial enrolling 78 patients with relapsed or refractory DLBCL.

DETAILED DESCRIPTION:
Participants will received 6 cycles every 21 days with a follow-up period of 24 months.

CT-Scan after 3 cycles and at the end of the treatment will be used to assess treatment response, established with Cheson criteria in 1999.

Principal objective is to obtain an overall response rate of 60% (corresponding to an increased of 15% of the rituximab-gemcitabine-oxaliplatine regimen's overall response rate).

Secondaries objectives are to value toxicity, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. patients from 18 to 75 years
2. Patient sharpened the social security system
3. Patients with relapsed or refractory diffuse large B cell lymphoma who received at least one prior line of immunochemotherapy unfit for intensive regimen therapy and autologous stem cell transplantation (ASCT) eligible patients to stem cell transplantation with failure of the salvage therapy patients with relapse after ASCT
4. Not previously treated with bendamustine
5. WHO performance status 0, 1 or 2
6. Adequate hematological function as defined by: leucocyte count ≥ 3.0 109/L, platelet count ≥ 75 109/L
7. Females of childbearing potential must agree to have a medically acceptable method of contraception from study treatment initiation until the end of treatment.
8. Signed informed consent.

Exclusion Criteria:

1. Person under guardianship or curatorship , or unable to understand the purpose of the study
2. Central nervous system or meningeal involvement
3. WHO performance status more than 2
4. Contraindication to any drug contained in the chemotherapy regimen
5. HIV disease, active hepatitis B or C
6. Any serious active disease or co-morbid medical condition
7. Any of the following laboratory abnormalities.

   * Leucocyte count < 3.0 x 109/L
   * Platelet count < 75 x 109/L
8. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
9. Pregnant or lactating females.
10. Prior history of malignancies, other than lymphoma, unless the patient has been free of the disease for ≥ 3 years. Exceptions include the following:

    * Basal cell carcinoma of the skin.
    * Squamous cell carcinoma of the skin.
    * Carcinoma in situ of the cervix.
    * Carcinoma in situ of the breast.
    * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b).
11. renal impairment with an estimated (modified dietin renal disease; MDRD) creatinine clearance < 40 ml/min,
12. chronic liver disease or day-1 (AST/ALT )≥2.5 upper limit of normal (ULN), total bilirubin≥1.5 ULN,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
treatment response | up to 20 weeks (at the end of the treatment)
  established with 1999 Cheson criteria on CT-scan

SECONDARY OUTCOMES:
overall survival | 2 years
progression free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gandhi Damaj, PHD, Study Director — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohmachi K, Niitsu N, Uchida T, Kim SJ, Ando K, Takahashi N, Takahashi N, Uike N, Eom HS, Chae YS, Terauchi T, Tateishi U, Tatsumi M, Kim WS, Tobinai K, Suh C, Ogura M. Multicenter phase II study of bendamustine plus rituximab in patients with relapsed or refractory diffuse large B-cell lymphoma. J Clin Oncol. 2013 Jun 10;31(17):2103-9. doi: 10.1200/JCO.2012.46.5203. Epub 2013 May 6. PMID 23650408
- [Background] Castegnaro S, Visco C, Chieregato K, Bernardi M, Albiero E, Zanon C, Madeo D, Rodeghiero F. Cytosine arabinoside potentiates the apoptotic effect of bendamustine on several B- and T-cell leukemia/lymphoma cells and cell lines. Leuk Lymphoma. 2012 Nov;53(11):2262-8. doi: 10.3109/10428194.2012.688200. Epub 2012 May 21. PMID 22530665
- [Background] Vacirca JL, Acs PI, Tabbara IA, Rosen PJ, Lee P, Lynam E. Bendamustine combined with rituximab for patients with relapsed or refractory diffuse large B cell lymphoma. Ann Hematol. 2014 Mar;93(3):403-9. doi: 10.1007/s00277-013-1879-x. Epub 2013 Aug 17. PMID 23955074
- [Background] Visco C, Finotto S, Pomponi F, Sartori R, Laveder F, Trentin L, Paolini R, Di Bona E, Ruggeri M, Rodeghiero F. The combination of rituximab, bendamustine, and cytarabine for heavily pretreated relapsed/refractory cytogenetically high-risk patients with chronic lymphocytic leukemia. Am J Hematol. 2013 Apr;88(4):289-93. doi: 10.1002/ajh.23391. Epub 2013 Feb 28. PMID 23450436
- [Background] Visco C, Finotto S, Zambello R, Paolini R, Menin A, Zanotti R, Zaja F, Semenzato G, Pizzolo G, D'Amore ES, Rodeghiero F. Combination of rituximab, bendamustine, and cytarabine for patients with mantle-cell non-Hodgkin lymphoma ineligible for intensive regimens or autologous transplantation. J Clin Oncol. 2013 Apr 10;31(11):1442-9. doi: 10.1200/JCO.2012.45.9842. Epub 2013 Feb 11. PMID 23401442
- [Result] Mounier N, El Gnaoui T, Tilly H, Canioni D, Sebban C, Casasnovas RO, Delarue R, Sonet A, Beaussart P, Petrella T, Castaigne S, Bologna S, Salles G, Rahmouni A, Gaulard P, Haioun C. Rituximab plus gemcitabine and oxaliplatin in patients with refractory/relapsed diffuse large B-cell lymphoma who are not candidates for high-dose therapy. A phase II Lymphoma Study Association trial. Haematologica. 2013 Nov;98(11):1726-31. doi: 10.3324/haematol.2013.090597. Epub 2013 Jun 10. PMID 23753028